CLINICAL TRIAL: NCT07161206
Title: The Effectiveness of a Digital Mindfulness Nudge Intervention on Well-Being, Cognitive, and Academic Outcomes in College Students: A Randomized Controlled Trial
Brief Title: The Effectiveness of a Digital Mindfulness Nudge Intervention on Well-Being, Cognitive, and Academic Outcomes in College Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Management University (Other)
Responsible Party: Principal Investigator, Tracy Chen Xi, Student, Singapore Management University PhD in Psychology, Singapore Management University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB-25-156-A124(825); C289 (Other Grant/Funding Number: Mrs Wong Kwok Leong Student Wellness Centre Fund)
Record Dates: First submitted 2025-08-25; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Digital Mindfulness Intervention
Keywords: Digital; Mindfulness; Nudge; Intervention; College Students

STUDY DESIGN:
Intervention Model Description: In the same duration, participants in the intervention/experimental group will be assigned to the intervention while participants in the control group will be assigned to a waitlist and receive no intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Mindfulness Intervention (Experimental): 28 Days of Daily Mindfulness Tasks
  Interventions: Behavioral: Digital Mindfulness Nudge Intervention
- Waitlist Control (No Intervention): Waitlist Control

INTERVENTIONS:
Behavioral: Digital Mindfulness Nudge Intervention — Participants will be guided through 28 Days of Mindfulness Exercises via a Telegram Channel (In a digital and nudge-based format)
  Arms: Digital Mindfulness Intervention

SUMMARY:
The goal of this controlled trial is to learn if a digital mindfulness nudge intervention named "28 Days of Mindful Moments" works to improve cognitive, well-being and academic outcomes in college students. The main questions it aims to answer are:

Cognitive: Does "28 Days of Mindful Moments" increase the level of mindfulness and decrease the level of rumination among participants? Well-Being: Does "28 Days of Mindful Moments" lower the levels of depression, anxiety, stress, negative affect and increase the levels of life satisfaction and positive affect among participants? Academic: Does "28 Days of Mindful Moments" increase the levels of productivity, study engagement, goal progress and decrease the levels of procrastination and study burnout among participants?

Researchers will compare the digital mindfulness nudge intervention to a waitlist control to see if the intervention works to improve the above outcomes.

Participants will:

Do daily mindfulness tasks/exercises such as mindful breathing or body scans for 1 month (28 Days) Fill in a questionnaire survey at two fixed time points (before and after for participants in the experimental group, before for participants in the control group) Fill in a follow-up survey

DETAILED DESCRIPTION:
The proposed study will be held as a collaboration between SMU Mrs Wong Kwok Leong Student Wellness Centre and SMU researchers. The study aims to examine the efficacy of a month-long Digital Mindfulness Nudge intervention on improving students' cognitive, academic and well-being outcomes.

The study utilises an experimental method of the experimental group filling in a survey (regarding cognitive, academic and well-being outcomes) before and after the intervention that they will be taking part in while the control group only fills in the surveys before they begin the intervention. Both the experimental group and the control group will fill in a baseline survey, before the experimental group begins their intervention. The intervention for the experimental group will last for 28 days. Meanwhile, the control group will be informed that due to an influx of participants, they can only start their intervention later. Another questionnaire survey will be sent to both the experimental and the control group to be filled in after the intervention ends for the experimental group. At this point, the experimental group would have completed the month-long mindfulness intervention while the control group would not have begun the intervention (i.e. they would have gone about their normal daily activities for the past month). The intervention will then take place for the control group. Additionally, to investigate longer term effects of the intervention, each of the conditions' (experimental and control) participants will also be encouraged to take part in a follow-up survey two weeks after their respective conditions, to see if any improvements in their cognitive, academic and well-being outcomes are long-lasting. The study is not intended to study the prevention, prognostication, diagnosis or alleviation of any disease, disorder or injury affecting the human body, such as psychological disorders.

ELIGIBILITY:
Inclusion Criteria:

* User of Telegram
* At least 18 years of age

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Mindful Attention Awareness | From enrollment to end of intervention (for experimental group) at the end of 28 Days and at Follow-up after 42 days.
  Mindful attention awareness will be measured using the 15-item Mindful Attention Awareness Scale MAAS (Brown & Ryan, 2003). Items like "I break or spill things because of carelessness" will be rated on a 6-point Likert scale from 1 (Almost always) to 6 (Almost never), where higher scores indicate greater mindfulness. Total scores will be computed by averaging item responses.

SECONDARY OUTCOMES:
Rumination | From enrollment to end of intervention (for experimental group) at the end of 28 Days and at Follow-up after 42 days.
  Rumination was measured using the 10-item Ruminative Responses Scale (Treynor et al., 2003), which assessed one's tendency to engage in repetitive and passive focus on symptoms of distress as well as their causes and consequences. Participants rate how frequently they engage in each response (e.g., "Think 'What am I doing to deserve this?'") on a 4-point Likert scale ranging from 1 (Never) to 4 (Always). Total scores will be computed by averaging the responses, with higher scores indicating greater rumination.
Depression | From enrollment to end of intervention (for experimental group) at the end of 28 Days and at Follow-up after 42 days.
  Depressive symptoms will be measured using the Centre of Epidemiologic Studies Depression Scale, 10-item revised version CES-D-R 10 (Andresen et al., 1994). Participants will respond to 10 items (e.g., "I felt that everything I did was an effort.") taking into account the past two weeks on a 4-point scale (1 = Rarely or none of the time, 4 = All of the time). Higher scores indicate higher levels of depressive symptomatology.
Anxiety | From enrollment to end of intervention (for experimental group) at the end of 28 Days and at Follow-up after 42 days.
  State anxiety will be assessed using the 6-item Spielberger State-Trait Anxiety Inventory STAI-6 (Marteau & Bekker, 1992). Six items (e.g., "I was tense these past 2 weeks.") will be rated from 1 (Not at all) to 4 (Very much so) and averaged for a composite score. Higher scores indicate greater levels of anxiety.
Stress | From enrollment to end of intervention (for experimental group) at the end of 28 Days and at Follow-up after 42 days.
  Stress will be evaluated using the 4-item Perceived Stress Scale PSS-4 (Cohen et al., 1983). Participants will rate items such as "How often have you felt difficulties piling up so high that you could not overcome them?" on a 0 to 4 scale (0 = Never to 4 = Very often). Higher scores indicate higher levels of perceived stress.
Positive affect | From enrollment to end of intervention (for experimental group) at the end of 28 Days and at Follow-up after 42 days.
  Positive affect will be measured using the Circumplex Model of Affect (Russell, 1980). Participants will rate feelings such as 'Pleasant', experienced over the past two weeks.
Negative Affect | From enrollment to end of intervention (for experimental group) at the end of 28 Days and at Follow-up after 42 days.
  Negative affect will be measured using the Circumplex Model of Affect (Russell, 1980). Participants rated feelings such as 'Irritable', experienced over the past two weeks.
Life Satisfaction | From enrollment to end of intervention (for experimental group) at the end of 28 Days and at Follow-up after 42 days.
  Life satisfaction will be measured using the Satisfaction with Life Scale (SWLS) (Diener et al., 1985). Participants will rate five items (e.g., "In most ways, these past 2 weeks have been close to ideal") on a 7-point scale (1 = Strongly disagree to 7 = Strongly agree). Scores will be averaged and higher scores will indicate higher life satisfaction.
Productivity | From enrollment to end of intervention (for experimental group) at the end of 28 Days and at Follow-up after 42 days.
  Productivity was assessed using five items drawn from the Task Performance subscale of the Individual Work Performance Questionnaire (IWPQ) (Koopmans et al., 2013; Koopmans et al., 2014). Participants will rate each item on a 0 to 5 scale (0 = Seldom, 5 = Always) for the past 2 weeks. Sample items include "I kept in mind the work result I needed to achieve" or "I managed my time well". The score will be computed as the mean of the five items, with higher scores indicating higher self-reported task performance.
Procrastination | From enrollment to end of intervention (for experimental group) at the end of 28 Days and at Follow-up after 42 days.
  Procrastination will be assessed using six items from the Irrational Procrastination Scale (Steel, 2002), such as "When I should be doing one thing, I did another." Participants will respond on a 1-5 scale, and higher scores indicate higher levels of procrastination.
Implementation intention and goal progress | From enrollment to end of intervention (for experimental group) at the end of 28 Days and at Follow-up after 42 days.
  Implementation Intention and Goal Progress were assessed using two face-valid items on a 5-point Likert scale (1 = Strongly disagree to 5 = Strongly agree). The implementation Intention question was "In the past 14 days, I have taken steps to achieve my goals for the month" while the goal progress question was "In the past 14 days, I have seen progress toward my goals for the month". Higher scores indicate greater implementation of intentions and greater progress toward monthly goals, respectively.
Study engagement | From enrollment to end of intervention (for experimental group) at the end of 28 Days and at Follow-up after 42 days.
  Study engagement will be measured using the 9-item Study Engagement Inventory (Salmela-Aro & Read, 2017), which measures students' energy, dedication, and absorption in their studies. Participants will rate items such as "When studying, I felt bursting with energy" based on their experiences over the past three weeks. Responses will be given on a 6-point Likert scale ranging from 1 (Completely disagree) to 6 (Completely agree). Higher scores indicate greater levels of academic engagement.
Study burnout | From enrollment to end of intervention (for experimental group) at the end of 28 Days and at Follow-up after 42 days.
  Study burnout will be measured using the 9-item Study Burnout Inventory (Salmela-Aro & Read, 2017), which assesses students' exhaustion, cynicism, and inadequacy in relation to their academic work. Participants will indicate how well each item describes their experiences over the past two weeks (e.g., "I felt overwhelmed by studying") on a 6-point Likert scale ranging from 1 (Completely disagree) to 6 (Completely agree). Scores were computed by averaging all items, with higher scores indicating greater academic burnout.

OTHER OUTCOMES:
Demographic outcomes | During baseline survey after enrollment
  Measures demographic characteristics such as age, sex, income, education etc
Data fidelity and intervention experience | From enrollment to end of intervention (for experimental group) at the end of 28 Days and at Follow-up after 42 days.
  Measured through a set of questions that ask about participants' motivation, honesty and satisfaction.

IPD SHARING:
Plan to Share IPD: No